CLINICAL TRIAL: NCT03916419
Title: A Single-Arm Phase II Study With a Safety Lead-in of Magnetic Resonance-Guided Hypofractionated Adaptive Radiation Therapy With Concurrent Chemotherapy and Consolidation Durvalumab for Inoperable Stage IIB, IIIA, and Select IIIB and IIIC Non-small Cell Lung Cancer
Brief Title: Magnetic Resonance-Guided Hypofractionated Adaptive Radiation Therapy With Concurrent Chemotherapy and Consolidation Durvalumab for Inoperable Stage IIB, IIIA, and Select IIIB and IIIC Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 201905035
Record Dates: First submitted 2019-04-12; First posted 2019-04-16 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Stage IIB Non-Small Cell Lung Cancer; Stage IIIA Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer; Stage IIIC Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy; Paclitaxel; Carboplatin; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Safety lead-in: Chemoradiation + Durvalumab (Experimental): * The first 6 patients enrolled on study will comprise the Safety Lead-In cohort and will be closely monitored for toxicity related specifically to the experimental chemoradiation portion of the study treatment. After these 6 patients have been enrolled, accrual will temporarily be suspended for a minimum of 6 months after completion of chemoradiation to allow for the evaluation of adverse events.
  * Patients will receive concurrent chemoradiation over the course of 3 weeks (15 fractions of radiation with online adaptive treatment planning at fractions 6, 9, and 12 and weekly carboplatin + paclitaxel). Four to 6 weeks after the end of chemoradiation, durvalumab immunotherapy will administered every 2 weeks or 4 weeks (timeline at the discretion of treating physician) for up to 12 months.
  Interventions: Device: ViewRay MR-Linear Accelerator; Radiation: Radiation therapy; Drug: Paclitaxel; Drug: Carboplatin AUC; Biological: Durvalumab
- Phase II: Chemoradiation + Durvalumab (Experimental): -Patients will receive concurrent chemoradiation over the course of 3 weeks (15 fractions of radiation with online adaptive treatment planning at fractions 6, 9, and 12 and weekly carboplatin + paclitaxel). Four to 6 weeks after the end of chemoradiation, durvalumab immunotherapy will administered every 2 weeks or 4 weeks (timeline at the discretion of the treating physician) for up to 12 months.
  Interventions: Device: ViewRay MR-Linear Accelerator; Radiation: Radiation therapy; Drug: Paclitaxel; Drug: Carboplatin AUC; Biological: Durvalumab

INTERVENTIONS:
Device: ViewRay MR-Linear Accelerator — -Radiation will be delivered by this machine
Radiation: Radiation therapy — -60Gy in 15 fractions
Drug: Paclitaxel — -50 mg/m^2 intravenous
  Other Names: Taxol
Drug: Carboplatin AUC — -2 mg/mL/min intravenous over 30 minutes
  Other Names: Paraplatin
Biological: Durvalumab — -10 mg/kg
  Other Names: Imfinzi

SUMMARY:
Building upon the clinical experience of the investigators with the magnetic resonance (MR)-guided radiation therapy system and applying principals of hypofractionation toward the current treatment paradigm of concurrent chemoradiation and consolidation immunotherapy for locally advanced non-small cell lung cancer (NSCLC), this prospective, single-arm Phase II clinical trial with safety lead-in will test the feasibility and outcomes of this approach.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven diagnosis of non-small cell lung cancer.
* Inoperable or patient has refused surgery
* Clinical AJCC stage IIB or IIIA (AJCC, 8th ed.) with plans to be treated with concurrent chemoradiotherapy.

  * Recurrent non-small cell lung cancer is allowed, provided the intent of the current treatment is curative and there has been no prior radiation to the thorax (except prior SBRT per the protocol)
  * Prior chemotherapy, immunotherapy, or targeted therapy is permitted as long as patients have recovered from prior toxicities to grade ≤ 1
  * Clinical AJCC stage IIIB with plans to be treated with concurrent chemoradiotherapy are eligible if any of the following apply: (1) T3N2M0, (2) T4N2M0 (with T4 by size criteria (> 7 cm); T4 due to invasion or nodules in other ipsilateral lobe are excluded), (3) T1-2N3M0 where N3 disease is confined to no more than 2 contiguous nodal stations in the contralateral mediastinum. N3 disease with either contralateral hilar adenopathy, multistation contralateral mediastinal adenopathy that is either non-contiguous or >2 contiguous nodal stations, or any scalene or supraclavicular adenopathy are not eligible.
  * Clinical AJCC stage IIIC (T3-4N3M0) are eligible if N3 disease is confined to no more than 2 contiguous nodal stations in the contralateral mediastinum as above and, if applicable, T4 is due only to size >7 cm as above.
* Appropriate stage for protocol entry based upon the following minimum diagnostic workup:

  * History/physical examination within 30 days prior to registration
  * FDG-PET/CT scan and CT chest with or without contrast for staging within 60 days prior to registration
  * MRI scan with contrast of the brain (preferred) or CT scan of the brain with contrast within 60 days prior to registration
* Zubrod Performance Status 0-2 within 30 days prior to registration.
* Age ≥ 18 years.
* CBC/differential obtained within 30 days prior to registration, with adequate bone marrow function defined as follows:

  * Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3
  * Platelets ≥ 100,000 cells/mm3
  * Hemoglobin ≥ 8.0 g/dl (Note: The use of transfusion or other intervention to achieve Hgb ≥ 8.0 g/dl is acceptable.)
* AST and ALT ≤ 1.5 upper limit of normal within 30 days prior to registration.
* Total bilirubin ≤ 1.5 upper limit of normal within 30 days prior to registration.
* Serum creatinine < 1.5 mg/dL or calculated creatinine clearance ≥ 50 mL/min within 30 days prior to registration estimated by the Cockcroft-Gault formula:

Creatinine Clearance (male) = [(140 - age) x (wt in kg)] [(Serum Creatinine mg/dl) x (72)] Creatinine Clearance (female) = 0.85 x Creatinine Clearance (male)

* Peripheral neuropathy ≤ grade 1 at the time of registration.
* Presence of measurable or evaluable disease by RECIST 1.1.
* Negative serum or urine pregnancy test within 2 weeks prior to registration for women of childbearing potential.
* Women of childbearing potential and male participants must agree to use a medically effective means of birth control throughout their participation in the treatment phase of the study.
* Able to understand and willing to sign an IRB-approved informed consent document. Patients without capacity to make an informed consent decision must have a legally authorized representative sign the IRB-approved informed consent document on their behalf.

Exclusion Criteria:

* Severe, active comorbidity, defined as follows:

  * Unstable angina, history of myocardial infarction and/or congestive heart failure requiring hospitalization within the last 6 months
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration;
  * Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for liver function and coagulation parameters are not required for entry into this protocol
  * Acquired Immune Deficiency Syndrome (AIDS) based upon current CDC definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive. Protocol-specific requirements may also exclude immuno-compromised patients
* Prior radiotherapy to the thorax. An exception can be made for prior stereotactic body radiation therapy (SBRT) if there is no overlap with the protocol PTV and OAR constraints can still be achieved with a composite plan.
* Evidence of a concurrent primary malignancy, or any history of metastatic cancer.
* Currently receiving any other investigational agents.
* Pregnant or breastfeeding.
* Medical contraindication to receiving MRI imaging (including presence of a cardiac pacemaker).
* Autoimmune disease requiring active treatment, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, or glomerulonephritis. Specific instances of autoimmune disease are eligible and allowed on study, as below:

  * Patients with a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone
  * Patients with controlled type 1 diabetes mellitus on a stable insulin regimen.
  * Patients with eczema or psoriasis with dermatologic manifestations only, provided that the disease is well controlled at baseline and only requiring topical steroids, with no acute exacerbations within the last 12 months (requiring psoralen, ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, high potency or oral steroids
* History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest CT scan.
* Chronic oral steroid use (greater than prednisone 10 mg orally once daily, or its equivalent) for any indication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2025-09-28 (Actual); Study Completion 2025-09-28 (Actual)

PRIMARY OUTCOMES:
Safety lead-in only: Number of participants with dose limiting toxicities (DLTs) | Through 6 months after completion of concurrent chemoradiation (estimated to be 6 months and 3 weeks)
  * Safety of hypofractionated MRI-guided adaptive radiotherapy (60Gy/15 fractions) with concurrent chemotherapy (carboplatin and paclitaxel) and consolidation durvalumab is defined as <2/6 participants experiencing dose limiting toxicities
  * DLT is defined as any possibly, probably, or definitely related to concurrent chemoradiation grade 3 toxicity that cannot be managed with maximal supportive care within 2 weeks, or any grade > 4 toxicity that occurs during treatment
  * The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be utilized for all toxicity reporting.
Local control rate (Phase II only) | Through 2 years after start of chemoradiation (estimated to be 2 years and 3 weeks)
  -Clinical and/or radiographic evidence of progression of disease at the primary (local) site
Regional control rate (Phase II only) | Through 2 years after start of chemoradiation (estimated to be 2 years and 3 weeks)
  -Clinical and/or radiographic evidence of progression of disease at the previously involved or uninvolved hilar and/or mediastinal nodal (regional) sites

SECONDARY OUTCOMES:
Number of acute toxicities | From start of chemoradiation through 60 days
  -Only those that are considered possibly/probably/definitely related to radiation therapy or chemoradiation
Number of late toxicities | From 61 days after start of chemoradiation through 2 years after the start of chemoradiation
  -Only those that are considered possibly/probably/definitely related to radiation therapy or chemoradiation
Tumor response rate | Through completion of treatment (estimated to be 12 months and 3 weeks)
  -Tumor response is defined as achieving a partial or complete response per RECIST criteria.
Distant recurrence rate | Through 2 years after start of chemoradiation (estimated to be 2 years and 3 weeks)
  -Distant recurrence is defined as development of metastatic, non-local, and non-regional disease.
Incidence of brain metastases | Through 2 years after start of chemoradiation (estimated to be 2 years and 3 weeks)
  -Defined as development of brain metastasis.
Progression-free survival (PFS) | Through 2 years after start of chemoradiation (estimated to be 2 years and 3 weeks)
  * Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).
  * PFS is defined as survival with no evidence of disease progression (local, regional, or distant) or death
Disease-free survival | Through 2 years after start of chemoradiation (estimated to be 2 years and 3 weeks)
  Disease-free survival is defined as survival with no evidence of recurrent (local, regional or distant) disease or death
Overall survival | Through 2 years after start of chemoradiation (estimated to be 2 years and 3 weeks)
  -Defined as survival with no evidence of death.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Vlacich, M.D, Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu